CLINICAL TRIAL: NCT05633160
Title: A Phase I/IIa Theranostic Study of 64Cu-SAR-BBN and 67Cu-SAR-BBN for Identification and Treatment of GRPR-expressing Metastatic Castrate Resistant Prostate Cancer in Patients Who Are Ineligible for Therapy With 177Lu-PSMA-617
Brief Title: 64Cu-SAR-BBN and 67CU SAR-BBN for Identification and Treatment of Gastrin Releasing Peptide Receptor (GRPR)-Expressing Metastatic Castrate Resistant Prostate Cancer in Patients Who Are Ineligible for Therapy With 177Lu-PSMA-617 (COMBAT)
Acronym: COMBAT
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Clarity Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLB05
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Prostatic Neoplasms; Castration-Resistant
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is to be conducted in 2 phases, a dose escalation phase and a cohort expansion phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 67Cu-SAR-BBN (Experimental): In the dose escalation phase:
  64Cu-SAR-BBN: Patients will receive up to 2 administrations of 200MBq
  67Cu-SAR-BBN: Cohorts 1 - 3: Single administration (dose will be determined based on cohort allocation).
  Cohort 4: 2 administrations at the recommended dose (determined by cohorts 1-3).
  In the cohort expansion phase:
  Patients will receive up to 3 administrations of 200MBq of 64Cu-SAR-BBN and 2 administrations at the recommended dose level of 67Cu-SAR-BBN, determined through the dose escalation.
  Additional administrations: (up to a maximum total of 4) may be offered to those participants, in either the dose escalation or cohort expansion, with radiological non-progression.
  Interventions: Drug: 64Cu-SAR-BBN; Drug: 67Cu-SAR-BBN

INTERVENTIONS:
Drug: 64Cu-SAR-BBN — 64Cu-SAR-BBN
Drug: 67Cu-SAR-BBN — 67Cu-SAR-BBN

SUMMARY:
The aim for this study is to determine the safety and efficacy of 67Cu-SAR-BBN in participants with Gastrin Releasing Peptide Receptor (GRPR)-expressing metastatic castrate resistant prostate cancer in patients who are ineligible for therapy with 177Lu-PSMA-617.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* ≥18 years of age;
* Eastern Cooperative Oncology Group performance status of 0 to 2;
* Life expectancy >6 months;
* Histological, pathological, and/or cytological confirmation of prostate cancer (PCa);
* ≥1 metastatic lesion that is present at screening computed tomography (CT), magnetic resonance imaging (MRI), or bone scan imaging obtained ≤28 days prior to enrollment into the study;
* Positive 64Cu-SAR-BBN PET/CT scan, where 64Cu-SAR-BBN uptake (standardized uptake value [SUV] max) of at least 1 known lesion is positive (higher than that of the liver). Any lesions on anatomical imaging larger in short axis than size as follows: organs ≥ 1 cm, lymph nodes ≥ 2.5 cm, bones (soft tissue component) ≥ 1 cm on the 1 hour positron emission tomography (PET)/ CT scan must also be positive for 64Cu-SAR-BBN uptake. NOTE: ALL OTHER ELIGIBILITY CRITERIA MUST BE FULFILLED BEFORE THE 64Cu-SAR-BBN ADMINISTRATION IS PERMITTED;
* Castrate level of serum/plasma testosterone (<50 ng/dL or <1.7 nmol/L);
* Have progressive mCRPC despite prior androgen deprivation therapy and at least either enzalutamide and/or abiraterone (or other such androgen receptor pathway inhibitors). Documented progressive mCRPC will be based on at least 1 of the following criteria:
* Serum/plasma prostate specific antigen (PSA) progression defined as 2 consecutive increases in PSA over a previous reference value measured at least 1 week prior. The minimal value for study enrollment is 2.0 ng/mL;
* Soft-tissue progression defined as a ≥20% increase in the sum of the diameter (SOD) (short axis for nodal lesions and long axis for non-nodal lesions) of all target lesions based on the smallest SOD since the last treatment directed at the metastatic cancer has started (not including hormonal therapy) or the appearance of 1 or more new lesions;
* Progression of bone disease: evaluable disease or new bone lesions(s) by bone scan.
* Participants must be ineligible for 177Lu-PSMA based therapy due to either of the following criterion:
* Participant is not a candidate for 177Lu-PSMA-based therapy in the opinion of the investigator, due to PET/CT characteristics predicting a poor response to therapy.
* Participant experienced disease progression or lack of response (post- or while on- 177Lu-PSMA-based therapy), as determined by clinical or radiological assessment.
* Participants must have recovered to ≤ Grade 2 from all clinically significant toxicities related to prior therapies (prior chemotherapy, radiation, immunotherapy, etc.);
* Participants must have adequate organ function:
* Bone marrow reserve:
* White blood cell (WBC) count ≥2.5 x 109/L (2.5 x 109/L is equivalent to 2.5 x 103/μL and 2.5 x K/μL and 2.5 x 103/cc and 2500/μL) OR
* Absolute neutrophil count (ANC) ≥1.5 x 109/L (1.5 x 109/L is equivalent to 1.5 x 103/μL and 1.5 x K/μL and 1.5 x 103/cc and 1500/μL);
* Platelets ≥100 x 109/L (100 x 109/L is equivalent to 100 x 103/μL and 100 x K/μL and 100 x 103/cc and 100,000/μL);
* Hemoglobin ≥9 g/dL (5.59 mmol/L);
* Total bilirubin ≤1.5 x the institutional upper limit of normal (ULN). For participants with known Gilbert's Syndrome ≤3 x ULN is permitted;
* Alanine aminotransferase or aspartate aminotransferase ≤3.0 x ULN OR ≤5.0 x ULN for participants with liver metastases;
* Estimated glomerular filtration rate (eGFR) ≥50 mL/min.
* For participants who are human immunodeficiency virus infected: Participant must be healthy and have a low risk of Acquired Immune Deficiency Syndrome related outcomes in the opinion of the Investigator;
* For participants who have partners of childbearing potential: Partner and/or participant must use a method of birth control with adequate barrier protection (as described in Section 5.4.3.1).

Exclusion Criteria:

* Major surgery within 12 weeks prior to enrollment into the study;
* Symptomatic brain metastasis;
* Histologic diagnosis that is predominantly small cell PCa;
* Prior history of leukemia or Myelodysplastic Syndrome;
* Diagnosis of Deep Vein Thrombosis or Pulmonary Embolism within 4 weeks prior to enrollment into the study;
* Unmanageable urinary tract obstruction;
* Evidence of progressive lesion(s) on MRI and/or CT (according to Response Evaluation Criteria in Solid Tumors V1.1) that is gastrin releasing peptide receptor (GRPR) negative on the 1 hour 64Cu-SAR-BBN PET/CT scan as determined at screening;
* Previous treatment with a systemic radionuclide, including:
* Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Actinium-225, Iodine-131 within 6 months or in case of Radium-223 within 3 months or in the case of 177Lu-PSMA-based therapy within 6 weeks of treatment initiation (Day 0), as long as the participant meets all safety eligibility criteria, and the nadir of toxicities has been reached, without prior approval of the medical monitor;
* Previous treatment with any systemic anti-cancer therapy (e.g., chemotherapy, immunotherapy or biological therapy [including monoclonal antibodies]) within 4 weeks prior to treatment on study with the exception of Luteinizing Hormone Releasing Hormone, any other androgen deprivation therapy (ADT) (if ADT is discontinued prior to enrolment, 14 days must elapse after abiraterone discontinuation and 28 days after enzalutamide before the participant can be enrolled) or low dose corticosteroids;
* Previous treatment with any investigational agents within 4 weeks prior enrollment into the study;
* Known hypersensitivity to the components of the investigational products or its analogues;
* Transfusion for the sole purpose of making a participant eligible for study inclusion;
* Spinal metastasis with symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression;
* Concurrent serious medical conditions, including, but not limited to, New York Heart Association class III or IV congestive heart failure, history of congenital prolonged QT syndrome, uncontrolled infection, known active hepatitis B or C, or other significant co-morbid conditions that in the opinion of the Investigator would impair study participation or cooperation;
* Diagnosed with other malignancies that are expected to alter life expectancy or may interfere with disease assessment. However, participants with a prior history of malignancy that has been adequately treated and who have been disease free for more than 3 years are eligible, as are participants with adequately treated non-melanoma skin cancer, superficial bladder cancer;
* Any condition or personal situation that would pose an unacceptable radiation safety risk (as per institution guidelines, state and/or national regulations) to the participant or care giver at the time of release following the completion of therapy (e.g., uncontrolled urinary incontinence, high dependency care);
* Participants in whom it is known that external beam radiotherapy is scheduled after enrollment into the study;
* Participants with QTc > 470 msec;
* Participants with persistent acute and/or chronic pancreatitis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or maximum feasible dose (MFD) of a single dose of 67Cu-SAR-BBN | Up to 8 weeks
  MTD as determined by cohort observations of dose limiting toxicities or MFD determined by the activity of the dose to be administered, when the MTD has not been reached.
Recommended dose of two doses of 67Cu-SAR-BBN | Up to 14 weeks
  Recommended dose as determined by cohort observations of dose limiting toxicities
Efficacy of 67Cu-SAR-BBN in terms of Prostate Specific Antigen (PSA) response | Up to 5 years
  Proportion of participants with ≥50% decline in PSA
Efficacy of 67Cu-SAR-BBN in terms of radiographic response | Up to 5 years
  Efficacy will be assessed via the overall response rate according to RECIST V1.1 for soft tissue disease and according to PCWG3 for bone lesions
Incidence of dose limiting toxicities [Safety and tolerability] of 67Cu-SAR-BBN | Up to 8 weeks
  Incidence of dose limiting toxicities following a single administration of 67Cu-SAR-BBN
Incidence of dose limiting toxicities [Safety and tolerability] of 67Cu-SAR-BBN | Up to 14 weeks
  Incidence of dose limiting toxicities following repeated administrations of 67Cu-SAR-BBN
Incidence of 67Cu-SAR-BBN treatment-emergent adverse events [Safety and tolerability] | Up to 12 months
  Adverse Events will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 5, following single or repeated administrations of 67Cu-SAR-BBN
Incidence of 67Cu-SAR-BBN adverse event of special interest [Safety and tolerability] | Up to 5 years
  Protocol defined adverse event of special interest following single or repeated administrations of 67Cu-SAR-BBN
Safety and tolerability of 67Cu-SAR-BBN: Number of Participants with changes from baseline in vital signs | Up to 24 weeks
  Change from baseline in vital signs following single or repeated administrations of 67Cu-SAR-BBN
Safety and tolerability of 67Cu-SAR-BBN: Number of Participants with changes from baseline in electrocardiogram (ECG) parameters | Up to 24 weeks
  Change from baseline in ECG parameters following single or repeated administrations 67Cu-SAR-BBN
Safety and tolerability of 67Cu-SAR-BBN: Number of Participants with changes from baseline in laboratory results | Up to 52 weeks
  Change from baseline in laboratory results following single or repeated administrations 67Cu-SAR-BBN
Incidence of 64Cu-SAR-BBN treatment-emergent adverse events [Safety and tolerability] | Up to 12 months
  Adverse Events will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 5, following single or repeated administrations of 64Cu-SAR-BBN

CONTACTS AND LOCATIONS:
Overall Officials: Clarity Pharmaceuticals, Study Director — Clarity Pharmaceuticals
Locations (6):
- United States (6):
  - Stanford University, Stanford, California
  - Biogenix Molecular, Miami, Florida
  - BAMF Health, Inc, Grand Rapids, Michigan
  - XCancer Omaha LLC, Omaha, Nebraska
  - Duke University, Durham, North Carolina
  - M D Anderson Cancer Centre, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taunk NK, Escorcia FE, Lewis JS, Bodei L. Radiopharmaceuticals for Cancer Diagnosis and Therapy: New Targets, New Therapies-Alpha-Emitters, Novel Targets. Cancer J. 2024 May-Jun 01;30(3):218-223. doi: 10.1097/PPO.0000000000000720. PMID 38753757